CLINICAL TRIAL: NCT00113555
Title: Clinical Investigation of an Adjustable Continence Therapy (ACT) Periurethral Prosthetic System for Treatment of Female Stress Urinary Incontinence With or Without Hypermobility
Brief Title: Adjustable Continence Therapy (ACT) Device for the Treatment of Female Stress Urinary Incontinence
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uromedica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URM01-01-01
Record Dates: First submitted 2005-06-08; First posted 2005-06-09 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Open Label Study, ACT (Adjustable Continence Therapy)
  Interventions: Device: ACT (Adjustable Continence Therapy)

INTERVENTIONS:
Device: ACT (Adjustable Continence Therapy) — surgically implanted device

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a minimally invasive surgical procedure in up to 160 implanted female patients in which two adjustable balloons (one on each side of the urethra) are implanted to treat urinary stress incontinence.

The results will be analyzed to demonstrate the effects of the device as well as its associated risks. Therapeutic success will be based on whether the patients demonstrate at least a one-grade (mean) reduction in the Stamey score at 12 months.

DETAILED DESCRIPTION:
This is a multi-center, prospective, non randomized clinical trial comparing baseline data to the 12 month data. Urodynamic testing, pad weights and a direct visual stress test will be used to determine success along with the Stamey score.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 years or older
* Diagnosed with stress urinary incontinence with or without urethral hypermobility
* Willing to sign informed consent
* Candidates for surgical intervention for stress incontinence
* Negative urinalysis or urine culture within 2 weeks of implantation
* Normal cystourethroscopy
* Failed at least 6 months of previous treatments for stress urinary incontinence (e.g., exercise regimen, electrical stimulation, surgical procedures, etc.)
* May have failed suspension or sling procedures

Exclusion Criteria:

* Pregnant or lactating
* Life expectancy of less than one year
* Insulin dependant diabetic
* Auto-immune disease
* Undergoing radiation therapy
* Active urinary tract infection
* Detrusor instability refractory to meds
* Reduced bladder compliance
* Significant bladder residual >100mls
* Bladder cancer
* Unsuccessfully treated bladder stones
* Current urethral stricture preventing the passage of a 24 French endoscope
* Neurogenic bladder
* Uncorrected rectocele, cystocele, urethrocele, enterocele or pelvic prolapse of Grade 3 or higher
* Prior pelvic radiotherapy
* Artificial urinary sphincter implanted

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2001-12; Primary Completion 2008-07 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Cook, Study Director — Uromedica, Inc.
Locations (7):
- United States (5):
  - Kaiser Permanente, Los Angeles, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Lahey Clinic, Burlington, Massachusetts
  - Metro Urology, Plymouth, Minnesota
  - Kansas City Urology Care, Kansas City, Missouri
- Canada (2):
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - CHUS-Fleurimont, Fleurimont, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 investigational sites in US and 2 in Canada which were clinics,University hospitals or Research centers implanted patients in this study from the period 2001-2006.A total of 221 patients have been enrolled(218 with enrollment data) and 163 of those patients underwent an implant procedure.
Pre-assignment Details: One patient was implanted and was considered a compassionate use patient that did not meet the enrollment criteria.This patient was not included in the efficacy and safety summaries and her adverse vents are recorded.Therefore the total number of implants for the analyses is 162.
Groups:
- ACT Adjustable Continence Therapy for Women: Open Label Study, patients implanted with ACT device for treatment of Stress Urinary Incontinence
Period: Overall Study
Arm/Group | ACT Adjustable Continence Therapy for Women
Started | 221
TREATED | 162 (1 Additional Patient was treated on a compassionate use basis.)
Completed | 142 (All treated patients were considered in the Intent to Treat analysis.)
Not Completed | 79
Not completed — Baseline Failure | 59
Not completed — Permanently Explanted | 7
Not completed — Death | 1
Not completed — Missed Followup | 4
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Open Label Study
Arm/Group | Experimental
Number analyzed (Participants) | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 137
  Canada | 25

OUTCOME MEASURES:

1. Primary Outcome: Change of Stamey Grade From Baseline to 12 Months.
Description: The Stamey grade classifies the severity of stress incontinence in four possible grades from 0-3. Grade 0: no leaking, Grade 1: loss of urine with sudden increases of abdominal pressure: e.g. coughing, sneezing or laughing, Grade 2: loss of urine with lesser degrees of stress: e.g. walking or standing up, and Grade 3: loss of urine without any relation to physical activity or position, e.g. while lying in bed.
  The primary end point at 12 months is a mean change in Stamey Grade from baseline of greater than or equal to -1.
Time Frame: Baseline to 12 months
Population: Intent to Treat
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 162
units on a scale | -1.17 [-1.33 to -1.01]
Statistical Analysis 1: Comparison: Experimental; Wilcoxon's matched pairs signed ranks test was used to determine the significance of differences between scores at follow-up compared to pre-implant; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -1.16, 95% CI 2-sided [-1.325 to -1.003], Standard Deviation 1.05

2. Secondary Outcome: Incontinence Quality of Life (IQoL) Questionnaire
Description: Change on Incontinence Quality of Life (IQoL) Questionnaire from baseline to 12 months. 0 being lowest quality of life, 100 being highest quality of life.
Time Frame: Baseline to 12 months
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ACT Adjustable Continence Therapy for Women: Open Label Study, patients implanted with ACT device for treatment of SUI
Arm/Group | ACT Adjustable Continence Therapy for Women
Number analyzed (Participants) | 162
units on a scale | 28.63 (29.69)

3. Secondary Outcome: Incontinence Impact Questionnaire (IIQ-7)
Description: Incontinence Impact Questionnaire (IIQ-7) change from baseline to 12 months. Scores range from 0-100. 0 being impact from incontinence, 100 being most impacted from incontinence.
Time Frame: Baseline to 12 months
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Adjustable Continence Therapy for Women
Number analyzed (Participants) | 162
units on a scale | -26.53 (33.07)

4. Secondary Outcome: Urinary Distress Inventory (UDI-6)
Description: Change on Urinary Distress Inventory (UDI-6) questionnaire from baseline to 12 months. 0 being not distressed, 100 being very distressed.
Time Frame: Baseline to 12 months
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Adjustable Continence Therapy for Women
Number analyzed (Participants) | 162
units on a scale | -22.66 (24.47)

5. Secondary Outcome: Number of Incontinence Episodes Per Day (Voiding Diary)
Description: Change in Number of Incontinence Episodes Per Day from baseline to 12 months. 0 being the best.
Time Frame: Baseline to 12 months
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT Adjustable Continence Therapy for Women
Number analyzed (Participants) | 162
units on a scale | -2.76 (5.06)

6. Secondary Outcome: Number of Pads Changed Per Day (Voiding Diary)
Description: Change in Number of Pads Changed Per Day from baseline to 12 months. 0 pads changed a day being the best.
Time Frame: Baseline to 12 months
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Number of Pads Changed per Day
Arm/Group | ACT Adjustable Continence Therapy for Women
Number analyzed (Participants) | 162
Number of Pads Changed per Day | -1.59 (3.63)

7. Secondary Outcome: Provocative Pad Weight
Description: Change in weight of pads (gm) from baseline to 12 months. 0 gm pad weight being the best.
Time Frame: Baseline to 12 months
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: gm
Arm/Group | ACT Adjustable Continence Therapy for Women
Number analyzed (Participants) | 162
gm | -31.03 (55.27)

ADVERSE EVENTS:
Time Frame: Entire Study December 2001 to November 2010 at Study Closure
Description: All adverse events were collected. Overall, although there were a large number of adverse events on the study (883) the majority were unrelated to the device (75%) or the procedure (82%) and 75% resolved with no residual effects. Of the 883 events, 270 of those events (31%) were considered device and/or procedure related.
Groups:
- ACT Adjustable Continence Therapy for Women: Open Label Study, Patients implanted with ACT device
Arm/Group | ACT Adjustable Continence Therapy for Women
All-Cause Mortality (participants affected / at risk) | 0/163
Serious Adverse Events (participants affected / at risk) | 2/163
Other Adverse Events (participants affected / at risk) | 155/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT Adjustable Continence Therapy for Women (N=163)
port erosion (Surgical and medical procedures) | 1 (1)
Other (non-pelvic) (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT Adjustable Continence Therapy for Women (N=163)
Pain/Discomfort (General disorders) | 51 (70)
Balloon Migration (General disorders) | 27 (32) — Balloon device moves from implantation site
Balloon Erosion (General disorders) | 10 (11) — Balloon Erodes into Vagina, Urethra, or Bladder
Port Migration (General disorders) | 7 (7) — Port moves from implantation site
Port Erosion (General disorders) | 21 (24) — Port erodes out of implantation site
Perforation (General disorders) | 14 (16) — Implantation tools perforate the vagina, urethra, or bladder during implantation procedure
Worsening Incontinence (Renal and urinary disorders) | 35 (37) — Patient has worsening incontinence symptoms
Device Failure (Product Issues) | 3 (4) — ACT device failure
Procedure Failure (General disorders) | 5 (5) — Procedure is not able to be completed
Infected Device (Infections and infestations) | 1 (1) — Infection of ACT Device
Other (Pelvic) (General disorders) | 75 (118)
Other (non-Pelvic) (General disorders) | 112 (336)
UTI (Renal and urinary disorders) | 75 (165) — Urinary Tract Infection
Yeast Infection (Renal and urinary disorders) | 21 (26)
Urinary Retention (Renal and urinary disorders) | 24 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No